CLINICAL TRIAL: NCT05467059
Title: Non-Interventional Study on Evaluation of Potential Causes of Nap Modulated Tinnitus
Brief Title: Evaluation of Potential Causes of Nap Modulated Tinnitus
Acronym: TinniNap
Status: Completed | Type: Observational
Sponsor: Robin Guillard EIRL (Industry)
Collaborators: Fondation Lopez-Loreta (Unknown); Service du sommeil de l'hôpital de l'Hôtel-Dieu (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-A00197-36
Record Dates: First submitted 2022-05-24; First posted 2022-07-20 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Tinnitus; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases
Keywords: Nap modulated tinnitus; Sleep modulated tinnitus; sleep apneas
MeSH Terms: conditions — Tinnitus; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nap-modulated participants: Patients with rises of tinnitus intensity after taking a nap or after a short period of sleep. If possible with a characteristic ON/OFF tinnitus (sometimes they have a tinnitus for several days and then stop for several days also). This condition is determined by previous questionnaire.
  Interventions: Other: Napping

INTERVENTIONS:
Other: Napping — Patients are already equipped with electrodes when they pass a test battery before the nap to evaluate mechanisms potentially correlated with tinnitus modulation. Then they do a nap, the nap is stopped when several periods of sleep are seen on EEG (electroencephalogram). Then the test battery is done backwards to evaluate the same measures.

SUMMARY:
The proposed research is a non-interventional study made to evaluate different measurements on 1 group of participants, before and after taking a nap, aiming to potentially guide future investigations on nap-modulated tinnitus to better understand this phenomenon.

The main hypothesis is that sleep apneas could be correlated with an increase of tinnitus intensity.

DETAILED DESCRIPTION:
1. - Background : Tinnitus is a really important concern due to its high prevalence (10% world population) and its deteriorating effects on life quality. Subjective tinnitus still remains a scientific enigma because of its partial elucidation. The limited knowledge on its causes can be partially attributed to its intrinsic heterogeneity. In questionnaires previous to this study, 34% of participants showed a characteristic symptomatology of interactions between tinnitus and their sleep : they feel their tinnitus at its maximum intensity after sleeping periods (nap and sleep). In most cases they describe a frank rise of the intensity, compared in scientific papers to the "exploding head syndrome". Therefore this study aims to determine what are the main physiopathological processes correlated to the rises of tinnitus
2. - Objectives : Estimate the correlations between tinnitus intensity changes (before and after the nap) and the number of sleep apneas. Secondary measurements are described in the outcome field.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated participant or beneficiary of a social security scheme
* Acceptation of protocol and signature of non-opposition
* Frankly nap-modulated tinnitus (increase of intensity after napping)
* Tinnitus maskable by white noise equal or inferior to 85 dB

Exclusion Criteria:

* Persons under juridic protection (guardianship or safeguard of justice)
* Clear cognitive incapacity (not understanding/nor apprehend the study tasks)
* Pregnancy or breast feeding
* Epilepsia
* Non-equilibrated chronic metabolic pathology
* Non-equilibrated psychiatric pathology
* Difficulty in napping
* Important hyperacusis
* Meniere's disease, fast fluctuating tinnitus (seconds or minutes), pulsatile tinnitus
* Any patient benefiting of a tinnitus treatment that was modified in the last 3 months
* Superficial wound, open or partially not cauterized

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is recruited through questionnaires done on different platforms including : SIOPI app, previous potential participants or associations. A lesser part of the study group comes from suggestions of ENTs/Doctors.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Average change in minimum masking level of tinnitus (measured in dB) | Average from 6 naps of 5 minutes sleep each over 2 days of participation
  Minimum masking level is measured with a wideband 20hz-12kHz noise before and after each nap of 5 minutes sleep.

SECONDARY OUTCOMES:
Correlation between sleep apnea index (number of apnea/hyponea events per hour) and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Sleep apnea index is measured during naps using plethysmography and using air flow measurements through cannulas.
Correlation between muscular tension (Electromyogram + Trigger Points) and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Using electromyogram on suprahyoid and masseter muscles, trigger points are done searching for muscle nodes
Correlation between Middle ear mobility (Impedancemetry) and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Using a multi-frequency impedancemeter
Correlation between tubal function (Tubomanometry) and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Using tubomanometer, the eustachian tube is controled (what pressure through the noise is needed)
Correlation between articular dysfunction (Physiotherapy Tests) and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Using cervical rotation test + adapted spurling test + jaw mobility in antepulsion and diduction
Correlation between change in averaged electroencephalogram alpha band power and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Difference of alpha band power in the EEG signal averaged on the whole scalp between the resting state of 90s before the 5 minutes nap and the one after.
Correlation between change in averaged electroencephalogram delta band power and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Difference of delta band power in the EEG signal averaged on the whole scalp between the resting state of 90s before the 5 minutes nap and the one after.
Correlation between change in averaged electroencephalogram theta band power and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Difference of theta band power in the EEG signal averaged on the whole scalp between the resting state of 90s before the 5 minutes nap and the one after.
Correlation between change in averaged electroencephalogram beta band power and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Difference of beta band power in the EEG signal averaged on the whole scalp between the resting state of 90s before the 5 minutes nap and the one after.
Correlation between change in averaged electroencephalogram gamma band power and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Difference of gamma band power in the EEG signal averaged on the whole scalp between the resting state of 90s before the 5 minutes nap and the one after.
Correlation coefficient between audition thresholds (Audiogram) values and change in minimum masking level of tinnitus (measured in dB) | 6 naps of 5 minutes sleep each over 2 days of participation
  Using an audiometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Hôtel-Dieu, Paris, France

IPD SHARING:
Plan to Share IPD: No